CLINICAL TRIAL: NCT01804153
Title: Phase II Clinical Trial to Study the Feasibility and Safety of the Expanded Autologous Mesenchymal Stem Cells Use Derived From Adipose Tissue (ASC) for the Local Feminine Stress Urinary Incontinence
Brief Title: Stem Cells Tratment for the Local Feminine Stress Urinary Incontinence Treatment (HULPURO)
Acronym: HULPURO
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HULPURO-2010-01; 2010-024331-16 (EudraCT Number)
Record Dates: First submitted 2012-09-04; First posted 2013-03-05 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Urinary Incontinence
Keywords: Feminine stress urinary incontinence; Autologous expanded stem cells
MeSH Terms: conditions — Urinary Incontinence

ARMS (1):
- Autologous expanded stem cells (Experimental): Adipose-derived expanded stem cells
  Interventions: Drug: Adipose-derived expanded stem cells

INTERVENTIONS:
Drug: Adipose-derived expanded stem cells — Intralesional application ASC

SUMMARY:
Evaluate the feasability and security of the autologous ASC for the femenine stress urinary incontinence

DETAILED DESCRIPTION:
Evaluate safety of adipose derived stem cells to femenine urinary incontinence with local application

ELIGIBILITY:
Inclusion Criteria:

1. -Signed informed consen
2. -Good general state of health according to the findings of ythe clinical history and the physical examination
3. -Postmenopausal or over 18 years old women taking highly effective contraceptives following the ICH (M3) EMA guide
4. -Women having rejected de rehabilitation treatment or in which the treatment had failed
5. -Genuine or combined stress urinary incontinence diagnosed with at least 1 year of evolution

Exclusion Criteria:

1. -Pregnant or lactating women
2. -Active urine infection
3. -Presenting an infravesical obstruction
4. -Alcohol or other addictive substances abuse antecedents in the previous 6 months to the inclusion
5. -Presenting any other malignant neoplasia unless it is a basocellar or a skin epidermoide carcinoma or presents antecedents of malignant tumours, unless they are in a remission phase for the previous 5 years
6. -Cardiopulmonar illness that, in the investigator opinion, could be unstable or could be serious enough to drop the patient from the study
7. -Any kind of medical or psychiatric illness that, in the investigator opinion, could be a reason to exclude the patient from the study
8. -Subjects with congenital or aquired inmunodeficiencies, B and/or C Hepatitis, Tuberculose or Treponema diagnosed at the moment of inclusion
9. -Anesthesic allergy
10. -Major surgery or severe trauma in the previous 6 months
11. -Administration of any drug under experimentation in the present or 3 months before recruitement

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-10 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Evaluate the feasability and security of the autologous ASC for the feminine stress urinary incontinence | 16 weeks
  compress test (number dthe changes daily) urethrocystoscopy (morphology of urethra)

SECONDARY OUTCOMES:
Quality of life assessment using the SF-12 Questionnaire | 1, 4, 16, 24 weeks
  SF-12 questionnaire
Adverse events | 1, 4, 16, 24 weeks
  Data collection

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Alonso Gregorio, MD, Principal Investigator — Hospital Universitario La Paz
Locations (1):
- Hospital Universitario La Paz, Madrid, Madrid, Spain

REFERENCES:
- [Background] Strasser H, Tiefenthaler M, Steinlechner M, Eder I, Bartsch G, Konwalinka G. Age dependent apoptosis and loss of rhabdosphincter cells. J Urol. 2000 Nov;164(5):1781-5. PMID 11025769
- [Background] Buckley BS, Lapitan MC; Epidemiology Committee of the Fourth International Consultation on Incontinence, Paris, 2008. Prevalence of urinary incontinence in men, women, and children--current evidence: findings of the Fourth International Consultation on Incontinence. Urology. 2010 Aug;76(2):265-70. doi: 10.1016/j.urology.2009.11.078. Epub 2010 Jun 11. PMID 20541241
- [Background] Mitterberger M, Pinggera GM, Marksteiner R, Margreiter E, Plattner R, Klima G, Strasser H. Functional and histological changes after myoblast injections in the porcine rhabdosphincter. Eur Urol. 2007 Dec;52(6):1736-43. doi: 10.1016/j.eururo.2007.05.007. Epub 2007 May 22. PMID 17532554
- [Background] Kwon D, Kim Y, Pruchnic R, Jankowski R, Usiene I, de Miguel F, Huard J, Chancellor MB. Periurethral cellular injection: comparison of muscle-derived progenitor cells and fibroblasts with regard to efficacy and tissue contractility in an animal model of stress urinary incontinence. Urology. 2006 Aug;68(2):449-54. doi: 10.1016/j.urology.2006.03.040. PMID 16904482
- [Background] Cannon TW, Lee JY, Somogyi G, Pruchnic R, Smith CP, Huard J, Chancellor MB. Improved sphincter contractility after allogenic muscle-derived progenitor cell injection into the denervated rat urethra. Urology. 2003 Nov;62(5):958-63. doi: 10.1016/s0090-4295(03)00679-4. PMID 14624934
- [Background] Praud C, Sebe P, Bierinx AS, Sebille A. Improvement of urethral sphincter deficiency in female rats following autologous skeletal muscle myoblasts grafting. Cell Transplant. 2007;16(7):741-9. doi: 10.3727/000000007783465118. PMID 18019363
- [Background] Becker C, Jakse G. Stem cells for regeneration of urological structures. Eur Urol. 2007 May;51(5):1217-28. doi: 10.1016/j.eururo.2007.01.029. Epub 2007 Jan 18. PMID 17254699
- [Background] Zuk PA, Zhu M, Mizuno H, Huang J, Futrell JW, Katz AJ, Benhaim P, Lorenz HP, Hedrick MH. Multilineage cells from human adipose tissue: implications for cell-based therapies. Tissue Eng. 2001 Apr;7(2):211-28. doi: 10.1089/107632701300062859. PMID 11304456
- [Background] Zhao W, Zhang C, Jin C, Zhang Z, Kong D, Xu W, Xiu Y. Periurethral injection of autologous adipose-derived stem cells with controlled-release nerve growth factor for the treatment of stress urinary incontinence in a rat model. Eur Urol. 2011 Jan;59(1):155-63. doi: 10.1016/j.eururo.2010.10.038. Epub 2010 Oct 26. PMID 21050657
- [Background] Kajbafzadeh AM, Elmi A, Payabvash S, Salmasi AH, Saeedi P, Mohamadkhani A, Sadeghi Z, Nikfarjam L. Transurethral autologous myoblast injection for treatment of urinary incontinence in children with classic bladder exstrophy. J Urol. 2008 Sep;180(3):1098-105. doi: 10.1016/j.juro.2008.05.057. Epub 2008 Jul 18. PMID 18639289
- [Background] Fu Q, Song XF, Liao GL, Deng CL, Cui L. Myoblasts differentiated from adipose-derived stem cells to treat stress urinary incontinence. Urology. 2010 Mar;75(3):718-23. doi: 10.1016/j.urology.2009.10.003. Epub 2009 Dec 6. PMID 19969332
- [Background] Lin G, Wang G, Banie L, Ning H, Shindel AW, Fandel TM, Lue TF, Lin CS. Treatment of stress urinary incontinence with adipose tissue-derived stem cells. Cytotherapy. 2010;12(1):88-95. doi: 10.3109/14653240903350265. PMID 19878076
- [Background] Carr LK, Steele D, Steele S, Wagner D, Pruchnic R, Jankowski R, Erickson J, Huard J, Chancellor MB. 1-year follow-up of autologous muscle-derived stem cell injection pilot study to treat stress urinary incontinence. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Jun;19(6):881-3. doi: 10.1007/s00192-007-0553-z. PMID 18204978
- [Background] Mitterberger M, Pinggera GM, Marksteiner R, Margreiter E, Fussenegger M, Frauscher F, Ulmer H, Hering S, Bartsch G, Strasser H. Adult stem cell therapy of female stress urinary incontinence. Eur Urol. 2008 Jan;53(1):169-75. doi: 10.1016/j.eururo.2007.07.026. Epub 2007 Jul 23. PMID 17683852
- [Background] Mitterberger M, Marksteiner R, Margreiter E, Pinggera GM, Colleselli D, Frauscher F, Ulmer H, Fussenegger M, Bartsch G, Strasser H. Autologous myoblasts and fibroblasts for female stress incontinence: a 1-year follow-up in 123 patients. BJU Int. 2007 Nov;100(5):1081-5. doi: 10.1111/j.1464-410X.2007.07119.x. Epub 2007 Aug 30. PMID 17760890
- [Background] Mitterberger M, Marksteiner R, Margreiter E, Pinggera GM, Frauscher F, Ulmer H, Fussenegger M, Bartsch G, Strasser H. Myoblast and fibroblast therapy for post-prostatectomy urinary incontinence: 1-year followup of 63 patients. J Urol. 2008 Jan;179(1):226-31. doi: 10.1016/j.juro.2007.08.154. Epub 2007 Nov 14. PMID 18001790
- [Background] Roche R, Festy F, Fritel X. Stem cells for stress urinary incontinence: the adipose promise. J Cell Mol Med. 2010 Jan;14(1-2):135-42. doi: 10.1111/j.1582-4934.2009.00915.x. Epub 2009 Oct 3. PMID 19799652
- [Background] Garcia-Olmo D, Garcia-Arranz M, Garcia LG, Cuellar ES, Blanco IF, Prianes LA, Montes JA, Pinto FL, Marcos DH, Garcia-Sancho L. Autologous stem cell transplantation for treatment of rectovaginal fistula in perianal Crohn's disease: a new cell-based therapy. Int J Colorectal Dis. 2003 Sep;18(5):451-4. doi: 10.1007/s00384-003-0490-3. Epub 2003 May 20. PMID 12756590
- [Background] Garcia-Olmo D, Herreros D, Pascual I, Pascual JA, Del-Valle E, Zorrilla J, De-La-Quintana P, Garcia-Arranz M, Pascual M. Expanded adipose-derived stem cells for the treatment of complex perianal fistula: a phase II clinical trial. Dis Colon Rectum. 2009 Jan;52(1):79-86. doi: 10.1007/DCR.0b013e3181973487. PMID 19273960